CLINICAL TRIAL: NCT05642520
Title: A Randomized Controlled Clinical Trial Comparing the Placement of an Oval Abutment in 2.9 mm Implants Versus a Circular Abutment in Implants of 3.3 mm to 12 Months of Evolution
Brief Title: Oval Abutment Versus a Circular Abutment in Dental Implants in the Anterior Maxillae
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ana María García de la Fuente (Other)
Responsible Party: Sponsor-Investigator, Ana María García de la Fuente, Professor, University of the Basque Country (UPV/EHU)
Organization: University of the Basque Country (UPV/EHU) (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2018_01
Record Dates: First submitted 2022-11-18; First posted 2022-12-08 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Dental Implants

STUDY DESIGN:
Intervention Model Description: The study was a double-blind controlled clinical trial (RCT) comparing the oval section abutment of a 2.9mm (test group) to a circular section abutment in 3.3mm (control group) implants for the replacement of a single tooth.
  The choice of the diameter to be used as recommended by the manufacter, was determined by the mesiodistal width between the two adjacent natural teeth, in order to maintain at least 1.5mm between the implant and the adjacent tooth. When said the distance was between 5.9 and 6.3 mm, a 2.9 mm implant was placed, while if the width ranged between 6.4 and 7.1 mm, a 3.3 mm implant was placed. Both implant designs are made of a titanium and zirconium alloy (Roxolid®) with a SLActive® surface (Institut Straumann AG, Basel, Switzerland).
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The clinical monitor will hide the treatment to the clinical observer, the patient and the statistician.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- oval section abutment of a 2.9mm (Experimental): The choice of the diameter to be used as recommended by the manufacter, was determined by the mesiodistal width between the two adjacent natural teeth, in order to maintain at least 1.5mm between the implant and the adjacent tooth. When said the distance was between 5.9 and 6.3 mm, a 2.9 mm implant was placed.
  Implant designs are made of a titanium and zirconium alloy (Roxolid®) with a SLActive® surface (Institut Straumann AG, Basel, Switzerland).
  Interventions: Procedure: Circular section abutment of 3.3 mm
- circular section abutment in 3.3mm (Placebo Comparator): The choice of the diameter to be used as recommended by the manufacter, was determined by the mesiodistal width between the two adjacent natural teeth, in order to maintain at least 1.5mm between the implant and the adjacent tooth. When said the distance was between 6.4 and 7.1 mm, a 3.3 mm implant was placed. Both implant designs are made of a titanium and zirconium alloy (Roxolid®) with a SLActive® surface (Institut Straumann AG, Basel, Switzerland).
  Interventions: Procedure: Oval section abutment of 2.9 mm

INTERVENTIONS:
Procedure: Oval section abutment of 2.9 mm — The choice of the diameter to be used as recommended by the manufacter, was determined by the mesiodistal width between the two adjacent natural teeth, in order to maintain at least 1.5mm between the implant and the adjacent tooth. When said the distance was between 5.9 and 6.3 mm, a 2.9 mm implant was placed. Implant designs are made of a titanium and zirconium alloy (Roxolid®) with a SLActive® surface (Institut Straumann AG, Basel, Switzerland).
  Arms: circular section abutment in 3.3mm
Procedure: Circular section abutment of 3.3 mm — The choice of the diameter to be used as recommended by the manufacter, was determined by the mesiodistal width between the two adjacent natural teeth, in order to maintain at least 1.5mm between the implant and the adjacent tooth. When said the distance was between 6.4 and 7.1 mm, a 3.3 mm implant was placed. Implant designs are made of a titanium and zirconium alloy (Roxolid®) with a SLActive® surface (Institut Straumann AG, Basel, Switzerland).
  Other Names: Prosthetic treatment over a circular section abutment of 3.3.mm
  Arms: oval section abutment of a 2.9mm

SUMMARY:
Objetive: The main objective of this clinical trial is to assess whether the oval section abutment of a 2.9mm implant achieves a greater covering of the tooth-implant papilla compared to a circular section abutment in 3.3mm implants in upper lateral incisors and lower central / lateral incisors.

Material and methods: fourty patients received unitary implants of 3.3mm or 2.9 mm diameter to replace the absence of upper lateral incisor or lower central/lateral incisor with an edentulous space of at least 6.4mm (mesio-distally). Esthetic and clinical parameters were evaluated 12 months after installation of the prosthesis.

Condition or disease: dental implants

Intervention/treatment: 3.3 or 2.9 mm diameter dental implants

Phase: Not Applicable

DETAILED DESCRIPTION:
The study was a double-blind controlled clinical trial (RCT) comparing the oval section abutment of a 2.9mm (test group) to a circular section abutment in 3.3mm (control group) implants for the replacement of a single tooth.

The choice of the diameter to be used as recommended by the manufacter, was determined by the mesiodistal width between the two adjacent natural teeth, in order to maintain at least 1.5mm between the implant and the adjacent tooth. When said the distance was between 5.9 and 6.3 mm, a 2.9 mm implant was placed, while if the width ranged between 6.4 and 7.1 mm, a 3.3 mm implant was placed. Both implant designs are made of a titanium and zirconium alloy (Roxolid®) with a SLActive® surface (Institut Straumann AG, Basel, Switzerland).

The main objective was the papillary index (PI) (Jemt, 1997). It consists in four scores: 0 = absence of interdental papilla; 1 = filling of the interdental space less than 50% of the soft tissues; 2 = filling of the interdental space greater than 50% of the soft tissues; 3 = total filling of the interdental space with good aesthetic harmony; 4 = Hyperplasic interdental papilla formation with irregular soft tissue. Both mesial and distal papilla will be recorded.

The secondary objectives are (a) to observe the stability of the soft and hard tissues after one year in function, (b) to assess the success and survival rate of the implants, (c) to assess the stability of the implants and their evolution and (d) to analyze the degree of patient satisfaction with the aesthetic result.

ELIGIBILITY:
Inclusion Criteria:

* Patients >18 years of age
* Absence of upper lateral incisors or lower central / lateral incisors with an edentulous space of at least 6.4mm (mesio-distally).
* The teeth adjacent to the edentulous space must be natural.
* Patients who are in periodontal health.
* Signing of informed consent before entering the study.

Exclusion Criteria:

* Patients with any systemic condition or disease that may interfere with oral surgery.
* History of radiotherapy.
* Patients smoking more than 20 cigarettes per day.
* Pregnant or breastfeeding patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
The main objective was the papillary index (PI) (Jemt, 1997) | 12 months
  It consists in four scores: 0 = absence of interdental papilla; 1 = filling of the interdental space less than 50% of the soft tissues; 2 = filling of the interdental space greater than 50% of the soft tissues; 3 = total filling of the interdental space with good aesthetic harmony; 4 = Hyperplasic interdental papilla formation with irregular soft tissue. Both mesial and distal papilla will be recorded.

SECONDARY OUTCOMES:
To observe the stability of the soft and hard tissues after one year in function: probing depth | 12 months
  Probing depth (PD), defined as the distance (mm) between the most apical point of the gingival sulcus or periodontal pocket and the free gingival margin. It will be taken at six points per tooth and in four points by implant.
To observe the stability of the soft and hard tissues after one year in function:bleeding on probing | 12 months
  Bleeding on probing (BP) (Ainamo and Bay 1975), presence of bleeding in six points per tooth (3 in vestibular and 3 in lingual or palatal).
To observe the stability of the soft and hard tissues after one year in function: suppuration on probing | 12 months
  Suppuration on probing, presence of pus within 15 seconds after probing.
To observe the stability of the soft and hard tissues after one year in function: Modified plaque index (MPI) | 12 months
  Modified plaque index (MPI) (Mombelli et al 1987): 0 = no plaque detected; 1 = detection of plaque when a periodontal probe passes over the surface of the implant; 2 = the plaque is visible to the naked eye; 3 = abundant plate.
Assessment of survival rate of the implants | 12 months
  The survival rate of the implants will be recorded taking into consideration Albrektsson et al.´s criteria. (Albrektson et al 1986)
Assessment of the success of the implants | 12 months
  The implant will be considered successful when: (a) non-detectable clinical mobility (manual test); (b) absence of radiolucency around the surface of the implant; (c) absence of persistent pain; (d) absence of recurrent peri-implant infection. (Buser et al. 1990)
Analyze the degree of patient satisfaction with the aesthetic result. | 12 months
  Visual analog scale (VAS): the general patient satisfaction will be evaluated. The specific satisfaction with respect to 5 parameters will also be recorded - aesthetics, mastication, phonation, comfort and self-esteem - using 10 cm visual analog scales calibrated with the terms "nothing satisfied" and "totally satisfied" at the left and right ends respectively.

CONTACTS AND LOCATIONS:
Overall Officials: ANA MARIA GARCIA DE LA FUENTE, PhD, Principal Investigator — University of the Basque Country (UPV/EHU)
Locations (1):
- Department of Stomatology II. UPV/EHU, Leioa, Biscay, Spain

IPD SHARING:
Plan to Share IPD: Yes
The data collected for the study will be identified by a code and only the researcher will be able to relate them. The personal data will be treated with absolute confidentiality in accordance with the Data Protection Law and will remain in the patient's clinical history. The coded data will only be used for the purposes of this project.
Supporting Information: SAP

REFERENCES:
- [Background] Klein MO, Schiegnitz E, Al-Nawas B. Systematic review on success of narrow-diameter dental implants. Int J Oral Maxillofac Implants. 2014;29 Suppl:43-54. doi: 10.11607/jomi.2014suppl.g1.3. PMID 24660189
- [Background] Patil RC, den Hartog L, van Heereveld C, Jagdale A, Dilbaghi A, Cune MS. Comparison of two different abutment designs on marginal bone loss and soft tissue development. Int J Oral Maxillofac Implants. 2014 May-Jun;29(3):675-81. doi: 10.11607/jomi.3363. PMID 24818207
- [Background] Froum SJ, Natour M, Cho SC, Yu PYC, Leung M. Expanded Clinical Applications of Narrow-Diameter Implants for Permanent Use. Int J Periodontics Restorative Dent. 2020 Jul/Aug;40(4):529-537. doi: 10.11607/prd.4565. PMID 32559035
- [Background] Roccuzzo A, Imber JC, Jensen SS. Need for lateral bone augmentation at two narrow-diameter implants: A prospective, controlled, clinical study. Clin Oral Implants Res. 2021 Apr;32(4):511-520. doi: 10.1111/clr.13721. Epub 2021 Mar 1. PMID 33548077
- [Background] Mombelli A, van Oosten MA, Schurch E Jr, Land NP. The microbiota associated with successful or failing osseointegrated titanium implants. Oral Microbiol Immunol. 1987 Dec;2(4):145-51. doi: 10.1111/j.1399-302x.1987.tb00298.x. No abstract available. PMID 3507627
- [Background] Ainamo J, Bay I. Problems and proposals for recording gingivitis and plaque. Int Dent J. 1975 Dec;25(4):229-35. PMID 1058834
- [Background] Buser D, Weber HP, Lang NP. Tissue integration of non-submerged implants. 1-year results of a prospective study with 100 ITI hollow-cylinder and hollow-screw implants. Clin Oral Implants Res. 1990 Dec;1(1):33-40. doi: 10.1034/j.1600-0501.1990.010105.x. PMID 2099210
- [Background] Albrektsson T, Zarb G, Worthington P, Eriksson AR. The long-term efficacy of currently used dental implants: a review and proposed criteria of success. Int J Oral Maxillofac Implants. 1986 Summer;1(1):11-25. No abstract available. PMID 3527955
- [Derived] Herrera-Perez P, Garcia-De-La-Fuente AM, Andia-Larrea E, Marichalar-Mendia X, Aguirre-Urizar JM, Aguirre-Zorzano LA. Clinical analysis of the tooth-implant papilla for two narrow-diameter titanium-zirconium implants in the anterior area: prospective controlled clinical study. BMC Oral Health. 2024 Mar 5;24(1):310. doi: 10.1186/s12903-024-04075-2. PMID 38443879